CLINICAL TRIAL: NCT04227678
Title: Postprandial Fatty Acid Metabolism in Subjects With Lipoprotein Lipase Deficiency
Acronym: AGL12
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, André Carpentier, tenured professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019-2764
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lipoprotein Lipase Deficiency
MeSH Terms: conditions — Hyperlipoproteinemia Type I | interventions — Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group- A0 (Other): Control group: Healthy subjects with fasting glucose < 5.6, 2-hour post 75g Oral Glucose Tolerance Test (OGTT) glucose < 7.8 mmol/l and HbA1c < 5.8%; fasting TG < 1.5 mmol/l);
  A0: without heparin administered
  Interventions: Dietary Supplement: liquid meal
- LPLD group-A0 (Other): LPLD group: LPL deficient subjects with history of fasting TG > 5 mmol/l and homozygote or compound heterozygote for a LPL-gene mutation;
  A0: without heparin administered
  Interventions: Dietary Supplement: liquid meal
- Control group-A1 (Other): Control group: Healthy subjects with fasting glucose < 5.6, 2-hour post 75g OGTT glucose < 7.8 mmol/l and HbA1c < 5.8%; fasting TG < 1.5 mmol/l);
  A1: with an intravenous (i.v.) heparin bolus (50 IU/kg i.v.) followed by 250 IU/h i.v. during 6 hours starting 15 minutes before ingestion of liquid meal.
  Interventions: Drug: Heparin; Dietary Supplement: liquid meal
- LPLD group-A1 (Other): LPLD group: LPL deficient subjects with history of fasting TG > 5 mmol/l and homozygote or compound heterozygote for a LPL-gene mutation;
  A1: with an intravenous (i.v.) heparin bolus (50 IU/kg i.v.) followed by 250 IU/h i.v. during 6 hours starting 15 minutes before ingestion of liquid meal.
  Interventions: Drug: Heparin; Dietary Supplement: liquid meal

INTERVENTIONS:
Drug: Heparin — an intravenous (i.v.) heparin bolus (50 IU/kg i.v.) followed by 250 IU/h i.v. during 6 hours, starting 15 minutes before ingestion of liquid meal
  Arms: Control group-A1; LPLD group-A1
Dietary Supplement: liquid meal — low fat meal: (500 mL, 898 Kcal, 13% fat, 20.3% protein and 62.3% carbohydrates) will be ingested over 20 minutes

SUMMARY:
Lipoprotein lipase (LPL) is an enzyme that plays an important role in removing triglycerides (TG) (molecules that transport dietary fat) from the blood. Patients with LPL deficiency (LPLD) display during their whole life very high plasma TG levels often associated with episodes of postprandial abdominal pain, malaise, blurred vision, dizziness (hyperchylomicronemia syndrome) that may lead to recurrent pancreatitis episodes. Because of their very slow clearance in blood of their chylomicron-TG, these patients need to severely restrict their dietary fat intake to avoid these complications. Fortunately, novel treatments are being developed to circumvent LPL deficiency (LPLD) metabolic effect on chylomicron-TG clearance. However, there is no data on how LPLD affect organ-specific dietary fatty acid metabolism nor how the novel therapeutic agents may change this metabolism. For example, it is currently not understood how subjects with LPLD store their DFA into adipose tissues and whether they are able to use DFA as a fuel to sustain their cardiac metabolism, as healthy individuals do. This study aims to better understand theses two questions.

DETAILED DESCRIPTION:
The study protocol includes 3 visits: the screening visit and 2 postprandial metabolic studies performed in random order at an interval of 7 to 14 days, and performed with (A1) and without (A0) an intravenous (i.v.) heparin bolus followed by 250 IU/h i.v during 6 hours. Each metabolic study will last 9 hours (with 6 hours postprandial) and will include PET and stable isotopic tracer methods. At time 0, a low fat liquid meal will be ingested over 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 8 healthy LPL-deficient individuals (LPLD subjects) with history of fasting TG > 5 mmol/l and homozygote or compound heterozygote for a LPL-gene mutation;
* 8 control subjects (fasting glucose < 5.6, 2-hour post 75g OGTT glucose < 7.8 mmol/l and HbA1c < 5.8%; fasting TG < 1.5 mmol/l);
* age 18 to 75 yo;
* To be willing and able to adhere to the specifications of the protocol;
* To have signed an informed consent document indicating that they understood the purpose

Exclusion Criteria:

* age < 18 yo;
* overt cardiovascular disease as assessed by medical history, physical exam, and abnormal ECG
* Treatment with a fibrate, thiazolidinedione, beta-blocker or other drug known to affect lipid or carbohydrate metabolism (except statins, metformin, and other antihypertensive agents that can be safely interrupted);
* Treatment with anti-hypertensive medication (only for LPL-deficient individuals);
* presence of liver or renal disease; uncontrolled thyroid disorder;
* previous diagnosis of heparin-induced thrombocytopenia;
* Treatment with oral anticoagulation medication or platelet aggregation inhibiting drugs;
* A history of major hemorrhagic event;
* smoking (>1 cigarette/day) and/or consumption of >2 alcoholic beverages per day;;
* Female of child-bearing potential who is pregnant, breast feeding or intends to become pregnant or pre-menopausal female with a positive serum pregnancy test at the time of enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Organ-specific Dietary Fatty Acid (DFA) partitioning | 2 months
  will be determined using oral administration of [18F ]-Fluoro-6-Thia- Heptadecanoic Acid (FTHA ) during whole-body acquisition.
Myocardial DFA uptake | 2 months
  will be assessed using oral administration of [18F]-FTHA during dynamic PET acquisition.

SECONDARY OUTCOMES:
Myocardial nonesterified fatty acids (NEFA) metabolism | 2 months
  will be determined using [11C]-palmitate during dynamic PET acquisition.
Dietary fatty acid oxidation rate | 6 months
  will be measured using breath [13C]-carbon dioxide enrichment
Total oxidation rate | 2 months
  will be determined by indirect calorimetry
postprandial plasma NEFA turnover | 6 months
  will be determined using stable isotope tracers of fatty acids
postprandial plasma glucose turnover | 6 months
  will be determined using stable isotope tracers of glucose
Left ventricular function by Positron Emitting Positron (PET) ventriculography | 2 months
  will be determined using [11C]-acetate PET/CT. 180 megabecquerel (MBq) will be administered by bolus injection
Myocardial oxidative metabolism | 2 months
  will be determined using i.v. [11C]-acetate during dynamic PET/CT scanning.
Insulin sensitivity | 6 months
  will be determined using a multiplex ELISA which will measure multiple analytes in a single experiment.
Liver nonesterified fatty acids (NEFA) metabolism | 2 months
  will be determined using [11C]-palmitate during dynamic PET acquisition.
Metabolites distribution in plasma | 2 months
  will be determined using oral administration of [18F]-FTHA

CONTACTS AND LOCATIONS:
Overall Officials: André Carpentier, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada